CLINICAL TRIAL: NCT00385008
Title: An Open Label, Single Dose, Parallel Group Study to Evaluate Absorption and Transit Characteristics of TREXIMA and RELPAX in Patients Inside and Outside of an Acute Migraine Attack.
Brief Title: TREXIMA and RELPAX Gastric Scintigraphy Inside and Outside a Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRX105848
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-08

CONDITIONS: Migraine Disorders
Keywords: Combination product, sumatriptan succinate, naproxen sodium, absorption, pharmacokinetics, disintegration, gastric transit, gastric scintigraphy
MeSH Terms: conditions — Migraine Disorders; Dental Caries | interventions — Sumatriptan; Naproxen; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other): open-label active drug
  Interventions: Drug: Combination Product (sumatriptan succinate / naproxen sodium)
- Arm 2 (Other): open-label active drug
  Interventions: Drug: RELPAX(eletriptan) 40mg Tablet

INTERVENTIONS:
Drug: Combination Product (sumatriptan succinate / naproxen sodium) — sumatriptan/naproxen sodium
  Arms: Arm 1
Drug: RELPAX(eletriptan) 40mg Tablet — eletriptan tablets
  Other Names: Combination Product (sumatriptan succinate / naproxen sodium)
  Arms: Arm 2

SUMMARY:
An evaluation of tablet disintegration and absorption and gastric transit of sumatriptan and naproxen sodium from a TREXIMA tablet and eletriptan from a RELPAX 40mg tablet.

ELIGIBILITY:
Inclusion Criteria:

* Consented males and nonpregnant females using adequate contraception, between 18 and 55 years of age, with at least 1-6 migraines per month for past 6 months. Subjects will be excluded for confirmed or suspected ischemic heart disease, uncontrolled hypertension at screening; a history of epilepsy or structural brain lesions which lowered the convulsive threshold; confirmed or suspected cardiovascular, cerebrovascular, peripheral vascular, congenital heart disease, or ischemic bowel disease; impaired hepatic or renal function; basilar or hemiplegic migraine. Other exclusion criteria included use of a monoamine oxidase inhibitor within 2 weeks before screening; ergot prophylactics in past 3 months; anticoagulants; smoking more than 10 cigarettes/day, evidence of alcohol or substance abuse; GI bleeding disorders, inflammatory bowel disease; or any concurrent medical or psychiatric condition that in the investigator's opinion could affect interpretation of efficacy or safety information or which otherwise contraindicated participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09-13 (Actual); Primary Completion 2006-11-24 (Actual); Study Completion 2006-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kori S, Byrd S, Doll W, Page R, and Sandefer E. Gastric Emptying and Absorption of a Sumatriptan with RT Technology 85mg and Naproxen Sodium 500mg Tablet. Cephalalgia 2007; Vol 27; 649.
- [Background] Kori S, Byrd S, Doll W, Page R, and Sandefer E. Gastroscintigraphic Evaluation of Gastric Emptying and Absorption of Another Conventionally Formulated Triptan. Cephalalgia 2007; Vol 27; 730.
- [Background] Kori S, Byrd SC, Doll WJ, Page RC, and Sandefer EP. Gastric Transit and Absorption of Sumatriptan and Naproxen from a Fixed Single-Tablet Sumatriptan RT Technology 85mg and Naproxen Sodium 500mg in Migraineurs both During and Outside a Migraine Attack: Evaluation by Gastric Scintigraphy. Headache 2007; 47(5):751.
- [Background] Kori S, Doll WJ, Page RC, Byrd SC, Sandefer EP. Gastric Transit and Absorption of Eletriptan, another Conventionally Formulated Triptan, in Migraineurs both During and Outside a Migraine Attack: Evaluation by Gastric Scintigraphy. Headache 2007; 47(5):752.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: TRX105848 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single site in the United States during 13 September 2006 to 24 November 2006. TREXIMA® tablet was a fixed dose combination of sumatriptan succinate 119 milligrams (mg) (equivalent to 85 mg of sumatriptan) and naproxen sodium 500 mg.
Pre-assignment Details: First ten participants enrolled received TREXIMA and the next ten enrolled received Relpax. In each group, the first 5 participants who had a migraine and who were able to attend the clinic received the extra dose of the respective treatment.
Groups:
- TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg): Ten participants received single dose of radio labeled TREXIMA tablet (fixed dose combination of sumatriptan succinate 119 mg [equivalent to 85 mg of sumatriptan] and naproxen sodium 500 mg), orally, in absence of migraine. Five participants out of these participants visited clinic when they were experiencing an acute migraine attack and received TREXIMA during migraine attack at clinic. Dosing was repeated up to 2 additional times for up to 4 total doses. Each treatment administration were separated by at least 7 days. Each dose was administered with 240 milliliter (mL) of water.
- Relpax (Eletriptan 40 mg): Ten participants received single dose of Relpax (eletriptan hydrobromide, 40 mg) tablet, orally, in absence of migraine. Five participants out of theses participants visited clinic when they were experiencing an acute migraine attack and received single dose Relpax (eletriptan hydrobromide, 40 mg) tablet during migraine attack at clinic. Dosing was repeated up to 2 additional times for up to 4 total doses. Each treatment administration were separated by at least 7 days. Each dose was administered with 240 mL of water.
Period: Overall Study
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
Started | 10 | 10
In Absence of Migraine | 10 | 10
In Presence of Migraine (5 participants out of 10 in each arm were re-dosed in presence of migraine.) | 5 | 5
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg): Ten participants received single dose of radio labeled TREXIMA tablet (fixed dose combination of sumatriptan succinate 119 mg [equivalent to 85 mg of sumatriptan] and naproxen sodium 500 mg), orally, in absence of migraine. Five participants out of these participants visited clinic when they were experiencing an acute migraine attack and received TREXIMA during migraine attack at clinic. Dosing was repeated up to 2 additional times for up to 4 total doses. Each treatment administration were separated by at least 7 days. Each dose was administered with 240 mL of water.
- Total: Total of all reporting groups
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.6 (7.50) | 33.3 (7.17) | 32 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to 10%, 50%, 90% and Complete Gastric Empting of the Radioactive Markers Representing Sumatriptan, Naproxen and Eletriptan
Description: Scintigraphic images were analyzed in a time-lapse format and regions of interest were drawn to include the stomach and small intestine. Images were recorded in a supine position and a series of 3 to 60 consecutive anterior scintigraphic images, each 1 minute in duration, were recorded using a clinical grade gamma camera. After this initial continuous imaging sequence, additional images were recorded to coincide with pharmacokinetic (PK) blood sampling times as necessary to monitor the tablet disintegration and transit time through the intestines. Prior to ingesting the radiolabeled dosage forms, two external markers (2-3 microcuries of indium-111 or technetium-99m) were placed on each participant to facilitate consistent positioning underneath the gamma camera. The first marker was placed on the right side of the participant's chest (approximately at the fifth intercostal rib) and a second marker was placed on the hip bone (approximately the left anterior superior ileac spine).
Time Frame: Day 1 of each treatment administration (For 30 days)
Population: Scintigraphy Population consisted of all participants with evaluable data from the scintigraphic images.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10 | 10
hours (hr)
  10% gastric emptying, Sumatriptan, Non-migraine: number analyzed (Participants) | 10 | 0
  10% gastric emptying, Sumatriptan, Non-migraine | 0.100 [0.03 to 0.62] |
  10% gastric emptying, Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  10% gastric emptying, Sumatriptan, Migraine | 0.130 [0.05 to 0.69] |
  10% gastric emptying, Naproxen, Non-migraine: number analyzed (Participants) | 10 | 0
  10% gastric emptying, Naproxen, Non-migraine | 1.195 [0.53 to 1.91] |
  10% gastric emptying, Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  10% gastric emptying, Naproxen, Migraine | 1.300 [0.85 to 2.73] |
  10% gastric emptying, Eletriptan, Non-migraine: number analyzed (Participants) | 0 | 10
  10% gastric emptying, Eletriptan, Non-migraine |  | 0.400 [0.00 to 0.62]
  10% gastric emptying, Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  10% gastric emptying, Eletriptan, Migraine |  | 0.410 [0.00 to 0.69]
  50% gastric emptying, Sumatriptan, Non-migraine: number analyzed (Participants) | 10 | 0
  50% gastric emptying, Sumatriptan, Non-migraine | 0.675 [0.13 to 1.80] |
  50% gastric emptying, Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  50% gastric emptying, Sumatriptan, Migraine | 1.070 [0.15 to 1.42] |
  50% gastric emptying, Naproxen, Non-migraine: number analyzed (Participants) | 10 | 0
  50% gastric emptying, Naproxen, Non-migraine | 2.260 [1.42 to 3.46] |
  50% gastric emptying, Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  50% gastric emptying, Naproxen, Migraine | 2.310 [1.39 to 4.38] |
  50% gastric emptying, Eletriptan, Non-migraine: number analyzed (Participants) | 0 | 10
  50% gastric emptying, Eletriptan, Non-migraine |  | 0.590 [0.02 to 2.57]
  50% gastric emptying, Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  50% gastric emptying, Eletriptan, Migraine |  | 0.890 [0.02 to 2.21]
  90% gastric emptying, Sumatriptan, Non-migraine: number analyzed (Participants) | 10 | 0
  90% gastric emptying, Sumatriptan, Non-migraine | 3.020 [2.00 to 4.29] |
  90% gastric emptying, Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  90% gastric emptying, Sumatriptan, Migraine | 3.440 [2.26 to 4.28] |
  90% gastric emptying, Naproxen, Non-migraine: number analyzed (Participants) | 10 | 0
  90% gastric emptying, Naproxen, Non-migraine | 4.290 [2.44 to 5.84] |
  90% gastric emptying, Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  90% gastric emptying, Naproxen, Migraine | 4.010 [2.81 to 8.75] |
  90% gastric emptying, Eletriptan, Non-migraine: number analyzed (Participants) | 0 | 10
  90% gastric emptying, Eletriptan, Non-migraine |  | 2.590 [0.03 to 4.48]
  90% gastric emptying, Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  90% gastric emptying, Eletriptan, Migraine |  | 2.490 [0.05 to 4.23]
  Complete gastric emptying,Sumatriptan,Non-migraine: number analyzed (Participants) | 10 | 0
  Complete gastric emptying,Sumatriptan,Non-migraine | 4.505 [2.50 to 6.06] |
  Complete gastric emptying, Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  Complete gastric emptying, Sumatriptan, Migraine | 4.000 [3.02 to 8.00] |
  Complete gastric emptying, Naproxen, Non-migraine: number analyzed (Participants) | 10 | 0
  Complete gastric emptying, Naproxen, Non-migraine | 4.760 [2.50 to 8.03] |
  Complete gastric emptying, Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  Complete gastric emptying, Naproxen, Migraine | 4.500 [3.52 to 9.97] |
  Complete gastric emptying, Eletriptan,Non-migraine: number analyzed (Participants) | 0 | 10
  Complete gastric emptying, Eletriptan,Non-migraine |  | 3.765 [0.20 to 10.02]
  Complete gastric emptying, Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  Complete gastric emptying, Eletriptan, Migraine |  | 3.510 [0.36 to 4.53]

2. Primary Outcome: Mean Area Under the Drug Concentration Time Curve (AUC) From Time of Dosing Through 2 Hour Post-dose [AUC (0-2)], Through 24 Hour [AUC (0-24)] and AUC From Time of Dosing Extrapolated to Infinity [AUC (0-inf)] for Sumatriptan and Naproxen
Description: Following TREXIMA administration, 6 mL blood sample was collected at pre-dose and then at 5, 10 , 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, and 75 minutes. Then at 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6 hour and at 8, 10, 12, 24, 48, 72 hour post-dose for each treatment administered. All available plasma supernatant was withdrawn from the precipitated blood fraction.
Time Frame: Pre-dose and then at 5 minute intervals through 60 minutes, at 75 minutes, every 30 minutes from 90 minutes through 6 hours, and at 8, 10, 12, 24, 48 and 72 hours post-dose for each treatment administered.
Population: PK parameter population comprised of all participants in the PK concentration population for whom PK parameters were calculated.
  PK concentration population comprised of all participants who had a sample obtained and analyzed. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hr per mL (µg*hr/mL)
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg)
Number analyzed (Participants) | 10
microgram*hr per mL (µg*hr/mL)
  AUC (0-24), Sumatriptan, Non-migraine | 231.526 (25.63)
  AUC (0-24), Sumatriptan, Migraine: number analyzed (Participants) | 5
  AUC (0-24), Sumatriptan, Migraine | 165.707 (38.05)
  AUC (0-inf), Sumatriptan, Non-migraine: number analyzed (Participants) | 9
  AUC (0-inf), Sumatriptan, Non-migraine | 231.999 (24.76)
  AUC (0-inf), Sumatriptan, Migraine: number analyzed (Participants) | 4
  AUC (0-inf), Sumatriptan, Migraine | 158.036 (41.67)
  AUC (0-2), Sumatriptan, Non-migraine | 65.156 (36.18)
  AUC (0-2), Sumatriptan, Migraine: number analyzed (Participants) | 5
  AUC (0-2), Sumatriptan, Migraine | 54.884 (22.28)
  AUC (0-24), Naproxen, Non-migraine | 570.54 (15.0)
  AUC (0-24), Naproxen, Migraine: number analyzed (Participants) | 5
  AUC (0-24), Naproxen, Migraine | 627.06 (20.6)
  AUC (0-inf), Naproxen, Non-migraine: number analyzed (Participants) | 9
  AUC (0-inf), Naproxen, Non-migraine | 901.13 (21.9)
  AUC (0-inf), Naproxen, Migraine: number analyzed (Participants) | 5
  AUC (0-inf), Naproxen, Migraine | 978.39 (23.4)
  AUC (0-2), Naproxen, Non-migraine | 23.16 (79.3)
  AUC (0-2), Naproxen, Migraine: number analyzed (Participants) | 5
  AUC (0-2), Naproxen, Migraine | 24.38 (117.5)

3. Primary Outcome: Mean AUC (0-inf) and AUC (0-2) for Eletriptan
Description: Following Relpax administration, 8 mL blood sample was collected at pre-dose and then at 5, 10 , 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, and 75 minutes. Then at 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6 hour and at 8, 10, 12 hour post-dose for each treatment administered. All available plasma supernatant was withdrawn from the precipitated blood fraction.
Time Frame: Pre-dose and then at 5 minute intervals through 60 minutes, at 75 minutes, every 30 minutes from 90 minutes through 6 hours, and at 8, 10, 12 hours post-dose for each treatment administered.
Population: The PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10
µg*hr/mL
  AUC (0-inf), Non-migraine: number analyzed (Participants) | 9
  AUC (0-inf), Non-migraine | 540.669 (78.75)
  AUC (0-inf), Migraine: number analyzed (Participants) | 5
  AUC (0-inf), Migraine | 570.860 (94.16)
  AUC (0-2), Non-migraine | 70.249 (97.29)
  AUC (0-2), Migraine: number analyzed (Participants) | 5
  AUC (0-2), Migraine | 78.092 (120.65)

4. Primary Outcome: Maximum Observed Drug Concentration (Cmax) for Sumatriptan and Naproxen
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The PK parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg)
Number analyzed (Participants) | 10
nanograms per milliliter (ng/mL)
  Sumatriptan, Non-migraine | 49.900 (33.00)
  Sumatriptan, Migraine: number analyzed (Participants) | 5
  Sumatriptan, Migraine | 45.676 (30.77)
  Naproxen, Non-migraine | 46.34 (25.5)
  Naproxen, Migraine: number analyzed (Participants) | 5
  Naproxen, Migraine | 56.36 (28.1)

5. Primary Outcome: Cmax for Eletriptan
Description: as for outcome 3
Time Frame: as for outcome 3
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10
ng/mL
  Non-migraine | 80.246 (61.19)
  Migraine: number analyzed (Participants) | 5
  Migraine | 91.323 (74.84)

6. Primary Outcome: Time of Maximal Drug Concentration (Tmax) for Sumatriptan and Naproxen
Description: as for outcome 2
Time Frame: as for outcome 2
Population: PK parameter Population
Measure: Median (Full Range); unit: hr
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg)
Number analyzed (Participants) | 10
hr
  Sumatriptan, Non-migraine | 2.000 [0.67 to 5.00]
  Sumatriptan, Migraine: number analyzed (Participants) | 5
  Sumatriptan, Migraine | 1.500 [0.33 to 4.50]
  Naproxen, Non-migraine | 4.50 [1.5 to 8.0]
  Naproxen, Migraine: number analyzed (Participants) | 5
  Naproxen, Migraine | 4.00 [1.5 to 10.0]

7. Primary Outcome: Tmax for Eletriptan
Description: as for outcome 3
Time Frame: as for outcome 3
Population: PK parameter Population
Measure: Median (Full Range); unit: hr
Arm/Group | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10
hr
  Non-migraine | 2.500 [0.83 to 6.00]
  Migraine: number analyzed (Participants) | 5
  Migraine | 2.000 [1.00 to 5.50]

8. Primary Outcome: Time to Complete Dispersion of the Sumatriptan and Naproxen Portions of the TREXIMA Tablet and of the Relpax Tablet
Description: Scintigraphic images were analyzed in a time-lapse format and regions of interest were to be drawn to include the stomach and small intestine. Images were recorded in a supine position and a series of 3 to 60 consecutive anterior scintigraphic images, each 1 minute in duration, were recorded using a clinical grade gamma camera. After this initial continuous imaging sequence, additional images were recorded to coincide with PK blood sampling times as necessary to monitor the tablet disintegration and transit time through the intestines. Prior to ingesting the radiolabeled dosage forms, two external markers (2-3 microcuries of indium-111 or technetium-99m) were placed on each participant to facilitate consistent positioning underneath the gamma camera. The first marker was placed on the right side of the participant's chest (approximately at the fifth intercostal rib) and a second marker was placed on the hip bone (approximately the left anterior superior ileac spine).
Time Frame: Day 1 of each treatment administered (For 30 days)
Population: Scintigraphy Population
Measure: Median (Full Range); unit: hr
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10 | 10
hr
  Sumatriptan, Non-migraine: number analyzed (Participants) | 10 | 0
  Sumatriptan, Non-migraine | 0.050 [0.05 to 0.25] |
  Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  Sumatriptan, Migraine | 0.050 [0.05 to 0.20] |
  Naproxen, Non-migraine: number analyzed (Participants) | 10 | 0
  Naproxen, Non-migraine | 1.125 [0.67 to 4.00] |
  Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  Naproxen, Migraine | 1.250 [1.00 to 3.00] |
  Eletriptan, Non-migraine: number analyzed (Participants) | 0 | 10
  Eletriptan, Non-migraine |  | 0.600 [0.05 to 0.83]
  Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  Eletriptan, Migraine |  | 0.670 [0.05 to 0.83]

9. Primary Outcome: Time to First Appearance of Sumatriptan, Naproxen and Eletriptan at the Proximal Small Intestine
Description: as for outcome 8
Time Frame: Day 1 of each treatment administered (For 30 days)
Population: Scintigraphy Population
Measure: Median (Full Range); unit: hr
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10 | 10
hr
  Sumatriptan, Non-migraine: number analyzed (Participants) | 10 | 0
  Sumatriptan, Non-migraine | 4.365 [2.46 to 7.01] |
  Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  Sumatriptan, Migraine | 4.350 [3.15 to 5.60] |
  Naproxen, Non-migraine: number analyzed (Participants) | 10 | 0
  Naproxen, Non-migraine | 4.510 [2.42 to 7.01] |
  Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  Naproxen, Migraine | 4.350 [4.19 to 6.40] |
  Eletriptan, Non-migraine: number analyzed (Participants) | 0 | 10
  Eletriptan, Non-migraine |  | 5.530 [3.73 to 12.00]
  Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  Eletriptan, Migraine |  | 5.810 [3.50 to 6.50]

10. Primary Outcome: Small Intestine Transit and Residence (Time to 50% Through Intestine) of the Radioactive Markers Representing Sumatriptan, Naproxen and Eletriptan
Description: as for outcome 8
Time Frame: Day 1 of each treatment administered (For 30 days)
Population: Scintigraphy Population
Measure: Median (Full Range); unit: hr
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10 | 10
hr
  Sumatriptan, Non-Migraine: number analyzed (Participants) | 10 | 0
  Sumatriptan, Non-Migraine | 2.895 [1.72 to 6.24] |
  Sumatriptan, Migraine: number analyzed (Participants) | 5 | 0
  Sumatriptan, Migraine | 2.990 [2.50 to 5.45] |
  Naproxen, Non-Migraine: number analyzed (Participants) | 10 | 0
  Naproxen, Non-Migraine | 2.550 [0.24 to 3.86] |
  Naproxen, Migraine: number analyzed (Participants) | 5 | 0
  Naproxen, Migraine | 2.230 [1.95 to 3.40] |
  Eletriptan, Non-Migraine: number analyzed (Participants) | 0 | 10
  Eletriptan, Non-Migraine |  | 4.335 [1.80 to 11.49]
  Eletriptan, Migraine: number analyzed (Participants) | 0 | 5
  Eletriptan, Migraine |  | 4.140 [2.13 to 6.25]

11. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to Day 30
Population: The Safety Population consisted of all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
Number analyzed (Participants) | 10 | 10
Participants
  Any AEs | 8 | 3
  Any SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and nSAEs were collected from start of the study treatment up to Day 30
Description: On treatment SAEs and nSAEs were reported for Safety Population.
Arm/Group | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) | Relpax (Eletriptan 40 mg)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TREXIMA (Sumatriptan 85 mg + Naproxen 500 mg) (N=10) | Relpax (Eletriptan 40 mg) (N=10)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dissociation (Psychiatric disorders) | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.